CLINICAL TRIAL: NCT07352280
Title: An Observational, Prospective, Real-World Study of Tislelizumab as Neoadjuvant Therapy for dMMR/MSI-H Stage II-III Colorectal Cancer
Brief Title: Neoadjuvant Therapy With Tislelizumab for dMMR/MSI-H Stage II-III Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5791
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colo-rectal Cancer (dMMR/MSI-H CRC)
Keywords: tislelizumab; dMMR/MSI-H stage II-III colorectal cancer; neoadjuvant therapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tumours
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- dMMR/MSI-H CRC: Patients with dMMR/MSI-H stage II-III colorectal cancer who received neoadjuvant treatment with tislelizumab

SUMMARY:
This study is a prospective, observational, real-world investigation. This study will evaluate the efficacy and safety of tislelizumab monotherapy before surgery in patients with mismatch repair deficient or microsatellite instability high (dMMR/MSI-H) locally advanced colorectal cancer.

All patients will receive three cycles of tislelizumab neoadjuvant therapy followed by curative surgery. Postoperatively, based on surgical pathology, patients will receive adjuvant therapy with a regimen selected by the investigator or adopt a watch-and-wait strategy. The investigators will conduct a 5-year prospective follow-up.

The investigators plan to enroll approximately 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, ECOG performance status score 0-2.
2. Pathologically confirmed stage II-III colorectal adenocarcinoma (according to AJCC 8th edition).
3. Histologically confirmed mismatch repair deficient or genetic testing confirmed microsatellite instability high tumor.
4. Signed written informed consent.

Exclusion Criteria:

1. The patient has a history of other serious conditions rendering them unsuitable for surgery.
2. Subjects with the following conditions: active autoimmune diseases, active infectious diseases, inflammatory bowel diseases; requiring long-term glucocorticoid or immunosuppressive therapy during treatment; history of immunodeficiency; history of organ transplantation or haematopoietic stem cell transplantation; severe interstitial pneumonia or pulmonary fibrosis.
3. Known hypersensitivity to any component or excipient of tislelizumab or other PD-1/PD-L1 agents.
4. Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal adenocarcinoma registered and treated at the Cancer Hospital Chinese Academy of Medical Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Up to 3 weeks after surgery
  The lack of all signs of cancer in tissue samples removed during surgery or biopsy after neoadjuvant treatment with tislelizumab.
Treatment emergent adverse events | Up to 90 days after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
  Treatment emergent adverse events (TEAE) are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment.

SECONDARY OUTCOMES:
Clinical complete response | Up to 6 weeks after 3 cycles (each cycle is 21 days) of neoadjuvant treatment
Event free survival | Up to 2 years
Overall survival | Up to 5 years
Treatment related adverse events | Up to 90 days after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment
Immunotherapy related adverse events | Up to 90 days after completion of 3 cycles (each cycle is 21 days) of neoadjuvant treatment